CLINICAL TRIAL: NCT01747330
Title: An Open Label, Multicenter Study Evaluating Safety and Tolerability of Creon Micro in Pediatric Subjects From at Least One Month to Less Than Four Years of Age With Pancreatic Exocrine Insufficiency Due to Cystic Fibrosis
Brief Title: Evaluation of Safety and Tolerability of Creon Micro in Children Younger Than Four Years With Pancreatic Exocrine Insufficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Products (Industry)
Responsible Party: Sponsor
Organization: Abbott (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M13-277
Record Dates: First submitted 2012-11-23; First posted 2012-12-11 (Estimated); Results first posted 2014-07-15 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-06

CONDITIONS: Pancreatic Exocrine Insufficiency
Keywords: cystic fibrosis
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Cystic Fibrosis | interventions — Pancreatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Creon micro, minimicrospheres (Experimental)
  Interventions: Drug: Pancreatin

INTERVENTIONS:
Drug: Pancreatin — Doses of Pancreatin <2500 lipase u/kg/feed or <4000 lipase U/g fat/intake or <10000 lipase U/kg/day given orally are used
  Other Names: Creon micro

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of Creon micro in children younger than four years with pancreatic exocrine insufficiency.

DETAILED DESCRIPTION:
A prospective open-label, multi-center study evaluating safety and tolerability of Creon Micro in pediatric subjects from at least one month to less than four years of age with Pancreatic Exocrine Insufficiency (PEI) due to Cystic Fibrosis (CF). Referring to the European Medicines Agency (EMEA) pediatric age criteria for the purpose of the study, subjects are categorized as infants and toddlers (< 2 years) and children, (2 years to < 4 years). In total, 40 subjects will be enrolled (20 subjects in each age subgroup). Subjects receive their prescribed pancreatic enzyme supplementation at the individual dose until start of treatment with Creon Micro, if the subjects were on pancreatic enzyme supplementation before start of the study. Subjects will be treated with Creon Micro during the study. The treatment duration is 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Children younger than four years with confirmed cystic fibrosis diagnosis and a body weight of at least 2 kilograms

Exclusion Criteria:

* Ileus or acute abdomen
* history of fibrosing colonopathy
* history of distal ileal obstruction without surgery
* solid organ transplant or surgery affecting the large bowel, other than appendectomy

Max Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suntje Sander-Struckmeier, PhD, Study Director — Abbott
Locations (9):
- Russia (9):
  - Site Reference ID/Investigator# 80716, Barnaul
  - Site Reference ID/Investigator# 80693, Moscow
  - Site Reference ID/Investigator# 80698, Novosibirsk
  - Site Reference ID/Investigator# 80713, Novosibirsk
  - Site Reference ID/Investigator# 80715, Orenburg
  - Site Reference ID/Investigator# 80694, Saint Petersburg
  - Site Reference ID/Investigator# 80714, Tomsk
  - Site Reference ID/Investigator# 80697, Voronezh
  - Site Reference ID/Investigator# 80696, Yaroslavl

REFERENCES:
- [Derived] Kashirskaya NY, Kapranov NI, Sander-Struckmeier S, Kovalev V. Safety and efficacy of Creon(R) micro in children with exocrine pancreatic insufficiency due to cystic fibrosis. J Cyst Fibros. 2015 Mar;14(2):275-81. doi: 10.1016/j.jcf.2014.07.006. Epub 2014 Jul 25. PMID 25066363

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Creon Micro, Minimicrospheres
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Creon Micro, Minimicrospheres
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.7 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 27
Region of Enrollment [Number; unit: participants]
  Russian Federation | 40

OUTCOME MEASURES:

1. Primary Outcome: Body Weight
Description: change from baseline at day 84
Time Frame: 3 months
Population: Full Analysis subject sample
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Creon Micro, Minimicrospheres
Number analyzed (Participants) | 40
kg | 0.75 (0.61)

2. Primary Outcome: Height
Description: change from baseline at day 84
Time Frame: 3 months
Population: Full Analysis subject sample
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Creon Micro, Minimicrospheres
Number analyzed (Participants) | 40
m | 0.026 (0.020)

3. Primary Outcome: Stool Frequency
Description: Average daily stool frequency during treatment period: Number of bowel movements per day
Time Frame: 3 months
Population: Full Analysis subject sample
Measure: Mean (Standard Deviation); unit: Bowel movements per day
Arm/Group | Creon Micro, Minimicrospheres
Number analyzed (Participants) | 40
Bowel movements per day | 2.1 (0.8)

4. Primary Outcome: Stool Consistency
Description: Assessment of stool consistency by the caregiver on a daily basis: hard, formed/normal, soft, watery
Time Frame: 3 months
Population: Full Analysis subject sample
Measure: Mean (Standard Deviation); unit: % of days with normal stool consistency
Arm/Group | Creon Micro, Minimicrospheres
Number analyzed (Participants) | 40
% of days with normal stool consistency | 55.4 (26.4)

5. Primary Outcome: Subject's Acceptance of Treatment
Description: Acceptance to Creon Micro. The caregiver should give his/her opinion based on the following scale: very good, good, moderate, and unsatisfactory.
Time Frame: 3 months
Population: Full Analysis subject sample
Measure: Number; unit: percentage of participants
Arm/Group | Creon Micro, Minimicrospheres
Number analyzed (Participants) | 40
percentage of participants
  very good | 37.5
  good | 52.5
  moderate | 10.0
  unsatisfactory | 0

6. Secondary Outcome: Number of Subjects With Adverse Events
Time Frame: 4 months
Population: Full Analysis subject sample
Measure: Number; unit: participants
Arm/Group | Creon Micro, Minimicrospheres
Number analyzed (Participants) | 40
participants | 16

7. Secondary Outcome: Pulse
Description: Change from Baseline at Day 84
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Creon Micro, Minimicrospheres
Number analyzed (Participants) | 40
bpm | -3.1 (9.4)

8. Secondary Outcome: Number of Participants With Findings During Physical Examination
Description: A physical examination was conducted by the physician. All abnormal findings were recorded as medical histories if present prior to start of study drug or as AEs otherwise. There was no separate documentation of physical examination findings in this study.
Time Frame: 3 months
Population: Full Analysis subject sample
Measure: Number; unit: participants
Arm/Group | Creon Micro, Minimicrospheres
Number analyzed (Participants) | 40
participants | 12

9. Secondary Outcome: Number of Participants With Clinical Relevant Safety Laboratory Values
Description: (hematology: hemoglobin, hematocrit, RBC count, WBC count, platelet count; biochemistry: glucose (fasting), creatinine, alkaline phosphatase, total bilirubin, ALAT (alanine amino transferase), ASAT (aspartate amino transferase), gamma-glutamyl transferase, uric acid, calcium, phosphate, potassium, serum pancreatic lipase; urinalysis (dipstick): glucose, blood, albumin, pH)
Time Frame: 3 months
Population: Full Analysis subject sample
Measure: Number; unit: participants
Arm/Group | Creon Micro, Minimicrospheres
Number analyzed (Participants) | 40
participants | 0

ADVERSE EVENTS:
Arm/Group | Creon Micro, Minimicrospheres
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 12/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Creon Micro, Minimicrospheres (N=40)
infections NEC (Infections and infestations) | 6 (8)
upper respiratory tract infections (Infections and infestations) | 3 (4)
gastrointestinal spastic and hypermotility disorders (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days